CLINICAL TRIAL: NCT05767359
Title: CAR- PRISM (PRecision Intervention Smoldering Myeloma): A Chimeric Antigen Receptor T Cell (CAR-T) Therapy Directed Against BCMA in High-Risk Smoldering Myeloma
Brief Title: CAR- PRISM (PRecision Intervention Smoldering Myeloma)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-546
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Smoldering Multiple Myeloma
Keywords: Multiple Myeloma; Smoldering Multiple Myeloma; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Cyclophosphamide; fludarabine phosphate; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Safety Run-In (Experimental): Participants will be enrolled into each of the 2 safety run-in phases in a standard 3 + 3 design.
  - Participants will undergo study procedures as outlined:
  * Apheresis for collection of peripheral blood mononuclear cells (PBMC) will occur on-site
  * Stem cell collection on-site post-apheresis per standard care.
  * Administration of Cyclophosphamide and fludarabine in pre-determined doses 1 x daily for 3 consecutive days.
  * Hospitalization to receive Cilta-cel in per-determined dose per protocol 1 x daily for 3 consecutive days and will remain in the hospital for 2 weeks post cilta-cell infusion.
  * Follow-up for 3 years post-treatment and up to 15 years.
  Interventions: Drug: Ciltacabtagene Autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate
- Cilta-Cel Dose Expansion Cohort (Experimental): Expansion cohort of 14 participants will be enrolled after safety run-in phases, and participants will undergo study procedures as outlined:
  * Apheresis for collection of peripheral blood mononuclear cells (PBMC) will occur on-site
  * Stem cell collection on-site post-apheresis per standard care.
  * Administration of Cyclophosphamide and fludarabine in pre-determined doses 1 x daily for 3 consecutive days.
  * Hospitalization to receive Cilta-cel in per-determined dose per protocol 1 x daily for 3 consecutive days and will remain in the hospital for 2 weeks post cilta-cell infusion.
  * Follow-up for 3 years post-treatment and up to 15 years.
  Interventions: Drug: Ciltacabtagene Autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate

INTERVENTIONS:
Drug: Ciltacabtagene Autoleucel — Genetically modified autologous T-cell immunotherapy, via intravenous infusion per protocol.
  Other Names: Cilta-cel, JNJ-68284528, LCAR-B38M
Drug: Cyclophosphamide — Lymphodepleting conditioning regimen, nitrogen mustard-derivative, via intravenous infusion per standard care.
  Other Names: Cytoxan
Drug: Fludarabine Phosphate — Lymphodepleting conditioning regimen, synthetic purine nucleoside, via intravenous infusion per standard care.
  Other Names: Fludarabine, Fludara

SUMMARY:
The goal of this research study is to test if ciltacabtagene autoleucel (cilta-cel) is safe and effective in treating participants with high-risk, smoldering myeloma.

The names of the treatment interventions used in this study are:

* Cilta-cel (or chimeric antigen receptor T cells)
* Cyclophosphamide (a lymphodepleting chemotherapy)
* Fludarabine (a lymphodepleting chemotherapy)

DETAILED DESCRIPTION:
This is a Phase II study to test the safety and effectiveness of study therapy cilta-cel in treating participants with high-risk smoldering multiple myeloma (SMM). T cells are a part of a person's immune system which usually helps fight infection and prevents/fights cancer cells.

The U.S. Food and Drug Administration (FDA) has approved cilta-cel as a treatment for relapsed and refractory multiple myeloma but not specifically for smoldering myeloma.

The research study procedures include screening for eligibility, study treatment including evaluations, blood collections, radiologic scans of tumors, bone marrow biopsies, and follow-up visits.

Participation in this study is expected to last about 15 years.

It is expected that about 20 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational therapy to learn whether the therapy works in treating a specific disease. "Investigational" means that the therapy is being studied.

Janssen Research & Development, LLC is supporting this research study by providing the study treatment and funding.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* High-risk SMM with ≤40% plasma cells in the bone marrow and with high-risk criteria defined as having 1 of the following 2 criteria:

  1. High-risk per "20-2-20" Criteria defined as presence of any two of the following:

     * Serum M-protein ≥ 2 gm/dL
     * Involved to uninvolved free light chain (FLC) ratio≥ 20
     * Bone marrow PC% ≥ 20% to <40%.
     * OR total score of 9 using the following scoring system:

       * FLC Ratio

         * >10-25 = 2
         * >25-40 = 3
         * > 40 = 5
       * Serum M-protein (g/dL)

         * >1.5-3 = 3
         * >3 = 4
       * BMPC%

         * >15-20 = 2
         * >20-30 = 3
         * >30-40 = 5
         * >40 = 6
       * FISH abnormality (t(4,14), t(14,16), 1q gain, or del13q = 2
  2. Presence of ≥10% BMPC and at least one of the following:

     * Evolving pattern:

       * eMP (≥10% increase in serum M-protein ) over a 6 month period OR;
       * Evolving change in hemoglobin (eHb) ≥ 0.5 g/dl decrease over a 12 months period OR;
       * Progressive Involved light chain increase >10% over a 6 month period along with a light chain ration > 8
     * Abnormal PC immunophenotype (≥95% of BMPCs are clonal) and reduction of ≥1 uninvolved immunoglobulin isotype. (Only IgG; IgA and IgM will be considered) High risk cytogenetics defined as presence of t(4;14), t(14;16), t(14;20), 17p deletion, TP53 mutation, 1q21 gain
* No evidence of CRAB criteria* or new criteria of active MM (SLIM-CRAB) which including the following:

  * Increased calcium levels: Corrected serum calcium >0.25 mmol/L (>1mg/dL) above the upper limit of normal or >2.75 mmol/L (>11mg/dL);
  * Renal insufficiency (attributable to myeloma);
  * Anemia (Hgb 2g/dL below the lower limit of normal or <10g/dL);
  * Bone lesions (lytic lesions or generalized osteoporosis with compression fractures)
  * No evidence of the following new criteria for active MM including the following:

    * Bone marrow plasma cells >60%
    * Serum involved/uninvolved FLC ratio ≥100
    * MRI with more than one focal lesion

      * Participants with CRAB criteria that are attributable to conditions other than the disease under study may be eligible after discussion with the Sponsor Investigator.
* ECOG Performance Status (PS) 0 or 1 (Appendix 8)
* The following laboratory values obtained < 28 days prior to registration:

  * ANC >1000/mL
  * PLT >75,000/mL
  * Total bilirubin ≤ 2.0 mg/dL (If total is elevated check direct and if normal patient is eligible.)
  * AST <2.5 x institutional upper limit of normal (ULN)
  * ALT <2.5 x institutional upper limit of normal (ULN)
  * Estimated creatinine clearance CrCl ≥60 mL/min (Cockcroft Gault equation).
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Women of childbearing potential must have a negative pregnancy test at screening.

  * When a woman is of childbearing potential, the following are required:

    • Subject must agree to practice a highly effective method of contraception (failure rate of <1% per year when used consistently and correctly) and agree to remain on a highly effective method of contraception from the time of signing the informed consent form (ICF) until 1 year after receiving a cilta-cel infusion. Examples of highly effective contraceptives include:
    * user-independent methods: 1) implantable progestogen-only hormone contraception associated with inhibition of ovulation; 2) intrauterine device; intrauterine hormone- releasing system; 3) vasectomized partner.
    * user-dependent methods: 1) combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral or intravaginal or transdermal; 2) progestogen-only hormone contraception associated with inhibition of ovulation (oral or injectable).
  * In addition to the highly effective method of contraception, a man:

    * Who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (eg, condom with spermicidal foam/gel/film/cream/suppository) from the time of signing the ICF until 1 year after receiving a cilta-cel infusion.
    * Who is sexually active with a woman who is pregnant must use a condom. Women and men must agree not to donate eggs (ova, oocytes) or sperm, respectively, during the study and for 1 year after the last dose of study treatment.

Note: Hormonal contraception may be susceptible to interaction with the study treatment, which may reduce the efficacy of the contraceptive method.

Exclusion Criteria:

* Prior SMM directed therapy.
* Symptomatic Multiple Myeloma or any evidence of CRAB criteria, including presence of myeloma defining events (MDE). Any prior therapy for active Myeloma should also be excluded. Bisphosphonates are not excluded.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational. Prior therapy with bisphosphonate is allowed. Prior radiation therapy to a solitary plasmacytoma is allowed but had to be at least 1 year prior to enrollment on the trial. Prior clinical trials or therapy for smoldering MM or MGUS are not allowed per exclusion criteria described above.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in-situ malignancy, or low-risk prostate cancer after curative therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, inflammatory disorders, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Plans to father a child while enrolled in this study or within 1 year after receiving the last dose of study drug.
* Pregnant or breast-feeding or planning to become pregnant while enrolled in this study or within 1 year after receiving the last dose of study drug.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) or SARS-CoV-2 (COVID-19).

  * Participants who are seropositive because of hepatitis B virus vaccine are eligible.
  * Participants who are positive for SARS-COV-2 antibody, HIV1 and 2 antibody, hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
  * Participants who are positive for HIV1 or 2 infections, with undetectable viral load and on stable antiretrovirals, will not be excluded.
  * Participants with past HCV infection that have now cleared will not be excluded.
* Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients (refer to Investigator's Brochure and appropriate package inserts).
* Prior or concurrent exposure to any of the following:

  1. Teclistamab, Belantamab, or any anti-BCMA therapy
  2. Investigational vaccine within 4 weeks of study therapy
  3. Live, attenuated vaccine within 4 weeks of study therapy.
  4. Monoclonal antibody therapy within 21 days except for those unrelated to MM therapy such as rituximab or other monoclonal antibodies for RA for example.
  5. Cytotoxic therapy within 14 days of study therapy
  6. PI therapy within 14 days of study therapy
  7. IMiD agent therapy within 14 days of study therapy
  8. Radiotherapy within 14 days or focal radiation within 7 days of study therapy.
* Known active CNS involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain MRI and lumbar cytology are required.
* Myelodysplastic syndrome or active malignancies (i.e., progressing or requiring treatment change in the last 24 months). The only allowed exceptions are:

  1. Non-muscle invasive bladder cancer treated within the last 24 months that is considered completely cured.
  2. Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured.
  3. Noninvasive cervical cancer treated within the last 24 months that is considered completely cured.
  4. Localized prostate cancer (N0M0):

     * With a Gleason score of <6, treated within the last 24 months, or untreated and under surveillance.
     * With a Gleason score of 3 or 4 that has been treated > 6months prior to study screening and considered to have a very low risk of occurrence, or
  5. History of localized prostate cancer and receiving androgen deprivation therapy and considered to have a very low risk of recurrence.
  6. Breast cancer: Adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer and receiving anti-hormonal agents and considered to have a very low risk of recurrence.
  7. Other malignancy that is considered cured with minimal risk of recurrence in the judgement of the investigator.
* Stroke or seizure within 6 months prior to signing ICF.
* Presence of the following cardiac conditions:

  1. New York Heart Association stage III or IV congestive heart failure
  2. Myocardial infarction or coronary artery bypass graft ≤6 months
  3. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
  4. History of severe non-ischemic cardiomyopathy
* Major surgery within 2 weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment.
* Concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study, such as:

  1. Uncontrolled diabetes.
  2. Acute diffuse infiltrative pulmonary disease.
  3. Evidence of active systemic viral, fungal, or bacterial infection, requiring systemic antimicrobial therapy.
  4. History of inflammatory disorders with the exception of vitiligo, type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing. Participants with mild rheumatoid arthritis will not be excluded.
  5. Disabling psychiatric conditions (e.g., alcohol or drug abuse), severe dementia, or altered mental status.
  6. Any other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
  7. History of non-compliance with recommended medical treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2040-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | 24 months
  Incidence of Dose Limiting Toxicities (DLTs) during the first 28 days after anti-BCMA CAR-T cell administration.
  Dose-Limiting Toxicities (DLTs) will be defined as follows:
  * Grade 4 non-hematologic toxicity of any duration including Grade 4 CRS and ICANS
  * Grade 3 CRS that does not improve to a grade 2 or less in 72 hours following adequate therapy.
  * Grade 3 neurological toxicity of any duration
  * Grade 3 toxicity of any duration involving vital organs (cardiac, pulmonary). Exceptions can be made if associated with CRS.
  * Other Grade 3 toxicity lasting > 72 hours. Exceptions may be made for Grade 3 abnormal hepatic or renal function tests that improve to grade 2 or less within 7 days.
  * Grade 3 hypersensitivity reaction that is not reversible to Grade 2 or less within 24 hours
  * Grade 4 neutropenia or thrombocytopenia lasting more than 28 days
Nature of Dose Limiting Toxicities (DLT) | 24 months
  Nature of Dose Limiting Toxicities (DLTs) during the first 28 days after anti-BCMA CAR-T cell administration.
  Dose-Limiting Toxicities (DLTs) will be defined as follows:
  * Grade 4 non-hematologic toxicity of any duration including Grade 4 CRS and ICANS
  * Grade 3 CRS that does not improve to a grade 2 or less in 72 hours following adequate therapy.
  * Grade 3 neurological toxicity of any duration
  * Grade 3 toxicity of any duration involving vital organs (cardiac, pulmonary). Exceptions can be made if associated with CRS.
  * Other Grade 3 toxicity lasting > 72 hours. Exceptions may be made for Grade 3 abnormal hepatic or renal function tests that improve to grade 2 or less within 7 days.
  * Grade 3 hypersensitivity reaction that is not reversible to Grade 2 or less within 24 hours
  * Grade 4 neutropenia or thrombocytopenia lasting more than 28 days
Incidence of Adverse Events (AEs) | 24 months
  Adverse events with onset or worsening on or after date of first dose of study treatment.
  AEs with onset or worsening on or after date of first dose of study treatment. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to AE. SAE is any untoward medical occurrence that results in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.

SECONDARY OUTCOMES:
Manufacture Success Rate (Feasibility) | 24 months
  Defined as number of subjects treated with planned target dose divided by total number of subjects treated, and it is done to evaluate the feasibility of the manufacturing process
Overall Response Rate (ORR) | 6 months
  Defined by the proportion of subjects with the best overall response (BOR). It is the BOR of stringent complete response (sCR), Complete response (CR), VGPR (Very good partial response), and Partial response (PR) at month 3 and month 6 as determined using International Myeloma Working Group (IMWG) Criteria (Kumar et al, 2016).
Complete Response Rate | 3 months
  Proportion of subjects with best overall response (BOR) of stringent complete response (sCR) or complete response (CR) at month 3 as determined by local investigator using International Myeloma Working Group (IMWG) Criteria (Kumar et al, 2016)
Duration of Response | 12 months from infusion of cellular product
  Duration of response (DOR) to be assessed, and DOR defined as the time from achievement of stringent complete response (sCR), Complete response (CR), VGPR (Very good partial response), and Partial response (PR) to relapse or death due to multiple myeloma.
Cmax of BCMA CAR-T Cells | 24 months
  Cmax of BCMA analyzed through qPCR-detected transgene of CAR-T concentrations over time in peripheral blood and bone marrow.
Tmax of BMCA CAR-T cells | 24 months
  Tmax of BCMA analyzed through qPCR-detected transgene of CAR-T concentrations over time in peripheral blood and bone marrow.
AUC of BCMA CAR-T cells | 24 months
  AUC of BCMA analyzed through qPCR-detected transgene of CAR-T concentrations over time in peripheral blood and bone marrow.
Clast of BCMA CAR-T cells | 24 months
  Clast of BCMA analyzed through qPCR-detected transgene of CAR-T concentrations over time in peripheral blood and bone marrow.
Number of patients with pre-existing and treatment induced immunogenicity of BMCA CAR-T | 24 months
  Both cellular and humoral of pre-existing and treatment induced immunogenicity for BCMA CAR-T cellular therapy in smoldering myeloma (SMM).

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu